CLINICAL TRIAL: NCT00467883
Title: AMBIZYGO: Efficacy of High Dose [10 mg/kg/j] Liposomal Amphotericin B (Ambisome)Efficacy in Initial Zygomycosis Treatment:Phase II Trial
Brief Title: Pilot Study of High Dose Liposomal Amphotericin B Efficacy in Initial Zygomycosis Treatment
Acronym: AMBIZYGO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P060603
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Zygomycosis
Keywords: Zygomycosis; High dose liposomal amphotericin B
MeSH Terms: conditions — Zygomycosis | interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- amphotericin B (Experimental): Treatment with high dosage of amphotericin B liposomal 10 mg/kg/day during 4 weeks
  Interventions: Drug: Liposomal Amphotericin B

INTERVENTIONS:
Drug: Liposomal Amphotericin B — high dosage
  Other Names: high dosage

SUMMARY:
Evaluation after 4 weeks of treatment or at end of treatment if it occurs before. Efficacy will be defined as objective responses; complete and partial response.

DETAILED DESCRIPTION:
Primary objective: Efficacy of 4 weeks of liposomal amphotericin B (AmBisome®) at high dose [10 mg/kg/j] or at maximal tolerable dose in initial zygomycosis treatment. Evaluation after 4 weeks of treatment or at end of treatment if it occurs before. Efficacy will be defined as objective responses; complete and partial response.

Secondary objectives: Efficacy, tolerance and survival after 15 days of treatment, cumulative dose of AmBisome® necessary to obtain objective response, efficacy in operated and non operated patients, tolerance after 4 and 12 weeks treatment, survival, and relapse rate at 6 months of 4 weeks of liposomal amphotericin B (AmBisome®) at high dose [10 mg/kg/j] or at maximal tolerable dose.

Scheme : prospective, multicentric, non comparative therapeutic pilot study.

Inclusion criteria: Presence on a tissue biopsy of large non septated hyphae compatible with zygomycete or presence of a zygomycete in culture associated with clinical or radiological abnormalities compatible with fungal invasive infection.

Exclusion criteria: Life expectancy below 72 hours, pregnancy, breast feeding, polyene hypersensitivity, absence of histologic or mycologic zygomycosis documentation, absence of informed consent, previous treatment with polyene or other antifungal active on zygomycete (posaconazole, itraconazole) over 5 days during the month previous inclusion.

Treatment : AmBisome® 10 mg/kg/j monotherapy during at least 15 days, then AmBisome® at maximal tolerable dose during 15 days associated with early optimal surgical treatment. After the first treatment month, following treatment is decided by referent physician.

ELIGIBILITY:
Inclusion Criteria:

* Presence on a tissue biopsy of large non septated hyphae compatible with zygomycete
* Presence of a zygomycete in culture associated with clinical or radiological abnormalities compatible with fungal invasive infection.

Exclusion Criteria:

* Life expectancy below 72 hours,
* Pregnancy, breast feeding,
* Polyene hypersensitivity,
* Absence of histologic or mycologic zygomycosis documentation,
* Absence of informed consent,
* Previous treatment with polyene or other antifungal active on zygomycete (posaconazole, itraconazole) over 5 days during the month previous inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2011-06 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Evaluation after 4 weeks of treatment or at end of treatment if it occurs before. Efficacy will be defined as objective responses; complete and partial response. | 4 weeks

SECONDARY OUTCOMES:
Efficacy, tolerance and survival after 15 days of treatment, cumulative dose of AmBisome® necessary to obtain objective response. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lortholary, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - Hôpital Necker - Service des Maladies Infectieuses et Tropicales, Paris
  - Necker Hospital, Paris

REFERENCES:
- [Derived] Lanternier F, Poiree S, Elie C, Garcia-Hermoso D, Bakouboula P, Sitbon K, Herbrecht R, Wolff M, Ribaud P, Lortholary O; French Mycosis Study Group. Prospective pilot study of high-dose (10 mg/kg/day) liposomal amphotericin B (L-AMB) for the initial treatment of mucormycosis. J Antimicrob Chemother. 2015 Nov;70(11):3116-23. doi: 10.1093/jac/dkv236. Epub 2015 Aug 27. PMID 26316385